CLINICAL TRIAL: NCT07244003
Title: Efficacy and Safety of the Triple Combination Therapy of Met/SGLT-2i/GLP-1RA or Other Oral Antidiabetic Drugs in Patients With Type 2 Diabetes Exhibiting Poor Glycemic Control
Brief Title: Efficacy and Safety of the Met+SGLT-2i+GLP-1RA in Patients With Type 2 Diabetes With Poor Glycemic Control
Acronym: MESSAGE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD-LLPHYJ-LC-1
Record Dates: First submitted 2025-11-16; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Liraglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Met+SGLT-2i+GLP-1RA (Experimental): Metformin+Ganagliflozin+Liraglutide
  Interventions: Drug: Metformin; Drug: ganagliflozin; Drug: liraglutide
- Triple Therapy of Other Oral Antidiabetic Drugs (Active Comparator): Building upon the previously stable treatment regimen, the addition of 1-2 oral hypoglycemic agents (excluding SGLT-2 inhibitors and oral GLP-1 receptor agonists) constitutes a triple oral hypoglycemic regimen.
  Interventions: Drug: Triple Therapy of Other Oral Antidiabetic Drugs

INTERVENTIONS:
Drug: Metformin — The dosage of metformin hydrochloride was consistent with baseline.
  Arms: Met+SGLT-2i+GLP-1RA
Drug: Triple Therapy of Other Oral Antidiabetic Drugs — The dosage of metformin hydrochloride was consistent with baseline. The usage and dosage of other hypoglycemic drugs were referred to their respective instructions.
  Arms: Triple Therapy of Other Oral Antidiabetic Drugs
Drug: ganagliflozin — Ganagliflozin tablet : 50mg/d.
  Arms: Met+SGLT-2i+GLP-1RA
Drug: liraglutide — Liraglutide injection: 0.6 mg/d for the first week, 1.2 mg/d for the second week, and 1.8 mg/d after the third week.
  Arms: Met+SGLT-2i+GLP-1RA

SUMMARY:
The main objective of this study is to compare the efficacy and safety of the triple combination therapy of Met/SGLT-2i/GLP-1RA or other oral antidiabetic drugs in patients with type 2 diabetes exhibiting poor glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for type 2 diabetes (refer to the Chinese Guidelines for the Prevention and Treatment of Type 2 Diabetes (2020 edition)); -Age: 18-75 years old (including the threshold), male or female;
* Body mass index (BMI) ≥20kg/m² ;
* Patients who took 1000mg or more of metformin in combination with or without another oral hypoglycemic agent (except SGLT-2i and oral GLP-1RA) for at least 8 weeks before screening and had poor blood glucose control (centralized detection of HBA1C >=7.5% and<=11.0%);
* Volunteer to participate in this study and sign informed consent.

Exclusion Criteria:

* Patients with type 1 diabetes or other special types of diabetes;
* Patients with acute complications of ketoacidosis/hyperglycemic hyperosmolar state/lactic acidosis within 6 months before screening
* Those who have used GLP-1RA and SGLT-2i drugs within 12 weeks before screening, or have used GLP-1RA and SGLT-2i drugs in the past and discontinued due to poor efficacy
* Those who received insulin treatment within the previous week
* Those who have a history of chronic or acute pancreatitis before screening, or have clinical manifestations of pancreatitis at the time of screening, or fasting triglycerides > 5.7 mmol/L during the screening period
* Liver function impairment at screening: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 UNL, or total blood bilirubin (TBIL) > 2 UNL;
* Renal impairment at screening: calculated according to the CKD-EPI formula, eGFR≤45 mL/min/1.73m² or serum creatinine≥1.5 UNL;
* Patients with a past or family history of medullary thyroid cancer (MTC) and patients with multiple endocrine neoplasia syndrome type 2 (MEN2)
* Female subjects who are currently pregnant, breastfeeding, or have a pregnancy plan during the study period
* Those who have a history of hypersensitivity reaction to metformin, gapagliflozin, liraglutide injection and other drugs used in research and their excipients or have contraindications to the study drugs;
* Those who have participated in other drug clinical trials within 3 months before screening; 21. Subjects who are unable to comply with the protocol under the judgment of the investigator, and those who have other serious physical or psychological diseases that may affect the effectiveness and safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-03-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The change of HbA1c compared to the baseline | from baseline to week 24

SECONDARY OUTCOMES:
The proportion of participants achieving HbA1c, blood pressure, and cholesterol targets | week 24
  HbA1c ≤ 7.0% Blood pressure < 130/80 mmHg For subjects without ASCVD, LDL-C < 2.6 mmol/L; for subjects with ASCVD, LDL-C < 1.8 mmol/L (< 70 mg/dL)
The proportion of patients achieving HbA1c target without hypoglycemia or weight gainning | week 24
  HbA1c target ≤ 7.0% The definition of hypoglycemia is: Blood glucose < 70 mg/dL ( < 3.9 mmol/L), regardless of whether there are symptoms of hypoglycemia.
The changes of waist circumference and hip circumference compared to the baseline | from baseline to week 24
The changes of fasting blood glucose, 2-hour post-meal blood glucose, fasting glucagon, fasting insulin, insulin resistance index (HOMA-IR) compared to the baseline | from baseline to week 24
Changes in systolic and diastolic blood pressure compared to the baseline | from baseline to week 24
The changes in urine albumin-to-creatinine ratio (UACR) compared to the baseline | from baseline to week 24
The changes of body mass compared to the baseline | from baseline to 24 week
The changes of BMI compared to the baseline | from baseline to 24 week
The changes of waist-hip ratio, waist-to-height ratio compared to the baseline | from baseline to 24 week

OTHER OUTCOMES:
The changes in total cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, alanine aminotransferase, and aspartate aminotransferase compared to the baseline | from baseline to week 120
The proportion of participants who received rescue treatment | from baseline to week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China